CLINICAL TRIAL: NCT01003652
Title: Harmonic Focus Shears Versus Clamp-and-technique for Total Thyroidectomy
Brief Title: Clinical Trial on Harmonic Focus Shears
Status: Completed | Type: Observational
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Other Study IDs: St Luc
Record Dates: First submitted 2009-10-27; First posted 2009-10-29 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Multinodular Goiter
Keywords: goiter
MeSH Terms: conditions — Goiter | interventions — Thyroidectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Harmonic Focus /conventional haemostasis
  Interventions: Procedure: thyroidectomy
- Harmonic Focus
- new surgical device
- Harmonic Focus / conventional haemostasis: Harmonic Focus group refers to the use of ultracision shears for haemostasis and conventional haemostasis group refers to the tie-and-clamp technique in total thyroidectomy

INTERVENTIONS:
Procedure: thyroidectomy — Comparison between two groups of patients. One group is operated on using harmonic Focus for haemostasis compared to a second group of patients operated on with the conventional haemostasis using tie-and-clamp technique
  Groups: Harmonic Focus /conventional haemostasis

SUMMARY:
The purpose of this study is to evaluate the technical benefits, advantages and limits of the use of the Harmonic Focus curved shears in total thyroidectomy.

DETAILED DESCRIPTION:
According to a randomized sequence, total thyroidectomy was performed in 34 patients using Harmonic Focus and in 34 patients using clamp-and-tie technique.

In this randomized prospective trial, differences in the duration of surgery, intraoperative bleeding and post-operative complications were analysed.

ELIGIBILITY:
Inclusion Criteria:

* Total thyroidectomy for multinodular goiter in adults patients

Exclusion Criteria:

* Redo surgery, malignancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 68 patients candidate to total thyroidectomy for multinodular goiter in an academic hospital
Sampling Method: Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2008-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Efficacy, safety and potential advantages of Harmonic Focus for total thyroidectomy | day one after surgery

SECONDARY OUTCOMES:
Impact on bleeding, operative time, instrument exchanges, material needed for haemostasis | during the operation

CONTACTS AND LOCATIONS:
Overall Officials: Michel Mourad, MD, PhD, Principal Investigator — St Luc
Locations (1):
- Cliniques universitaires Saint-Luc- Université Catholique de Louvain, Brussels, Belgium